CLINICAL TRIAL: NCT07244016
Title: Clinical Study on Using T Cell Repertoire Technology to Predict the Therapeutic Effect of Tislelizumab + Standard Chemotherapy in the First-line Treatment of Extensive-stage Small Cell Lung Cancer
Brief Title: Clinical Study on Using TCR to Predict the Effect of Tislelizumab + Chemotherapy in the First-line Treatment of ES-SCLC
Acronym: ES-SCLC
Status: Recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HXNY-TI-001
Record Dates: First submitted 2025-05-08; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-02

CONDITIONS: Extensive-stage Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational clinical study designed to predict the therapeutic efficacy of first-line treatment with tislelizumab combined with standard chemotherapy in patients with ES-SCLC using TCR repertoire technology. The study plans to enroll 40 treatment-naive patients with ES-SCLC.

DETAILED DESCRIPTION:
The advancement of Next-Generation Sequencing (NGS) technology has facilitated the detection of T-cell immune repertoires across various solid tumor types, and a growing body of research indicates that T-cell immune repertoires hold potential as biomarkers for immunotherapy; in the field of non-small cell lung cancer (NSCLC), previous studies have suggested that the characteristics of the baseline T-cell receptor (TCR) repertoire and changes in the TCR repertoire before and after immunotherapy are associated with immunotherapeutic efficacy, while such exploration remains lacking in the field of small cell lung cancer (SCLC). Due to limitations in cost and experimental methods, the currently available TCR databases contain limited information, encompassing only a small fraction of antigen-TCR binding pairs, and furthermore, these binding pair data fail to cover all antigens that any given TCR might potentially bind to; to address this issue, the research community has explored the use of machine learning models to predict the antigen specificity of unknown and experimentally unvalidated TCRs, which has shown feasibility. This study, as a prospective observational clinical study designed to predict the therapeutic efficacy of first-line treatment with tislelizumab combined with standard chemotherapy in patients with extensive-stage small cell lung cancer (ES-SCLC) using TCR repertoire technology, plans to enroll 40 treatment-naive patients with ES-SCLC, and aims to predict the neoantigen-specific TCR repertoire by analyzing tumor neoantigens, integrating T-cell repertoire data and HLA class I detection information, and leveraging the Multimodal-AIR-BERT machine learning model, with the hypothesis that the parameters of this predicted TCR repertoire may exhibit a stronger correlation with immunotherapeutic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven ES-SCLC (American Joint Cancer Commission (7th Edition) Stage IV SCLC [any T, any N and M1a/b]), or T3-4 patients who are unable to be included in a tolerable radiotherapy program due to wide multiple incidences or excessive tumor volume.
* Patients with brain metastases must have asymptomatic or stable steroid and anticonvulsant treatment for at least 1 month before study treatment. Patients with suspected brain metastasis during screening should undergo brain CT/MRI examination before enrollment of the study.
* Have at least one measurable tumour lesion according to RECIST v1.1.
* aged ≥18 years
* Eastern Cooperative Oncology Group (ECOG) physical status score of 0-1

Exclusion Criteria:

* Have a history of chest radiotherapy or plan to undergo intensive chest radiotherapy before systemic treatment. Radiotherapy outside the chest (i.e., bone metastasis) is allowed for palliative care purposes, however, must be done before the first medication of the study drug
* Previous non-infectious pneumonia requiring systemic glucocorticoid therapy or current non-infectious pneumonia combined with mild to moderate interstitial pneumonia, inactive interstitial pneumonia.
* Presence of unmitigated toxicity from prior antineoplastic therapy, with unmitigated defined as failure to recover to NCI CTCAE version 5.0 grade 0 or 1 (except alopecia areata) or failure to recover to levels specified in the inclusion/exclusion criteria.
* History of known allogeneic organ transplantation and allogeneic haematopoietic stem cell transplantation; history of organ or haematopoietic stem cell transplantation requiring immunosuppression.
* Patients with chronic hepatitis B or chronic hepatitis B virus carriers with HBV DNA ≥500 IU/mL (2500 copies/mL), or hepatitis C patients.
* Other circumstances as determined by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven ES-SCLC (American Joint Cancer Commission (7th Edition) Stage IV SCLC [any T, any N and M1a/b]), or T3-4 patients who are unable to be included in a tolerable radiotherapy program due to wide multiple incidences or excessive tumor volume.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival time | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from enrollment to either radiological progression or death

CONTACTS AND LOCATIONS:
Overall Officials: Chen Li Juan, Prof, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hosipital, Zhengzhou, Henan, China